CLINICAL TRIAL: NCT00332982
Title: Ontario ICU Clinical Best Practices Demonstration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Huntsville District Memorial Hospital (Unknown); Lake Of The Woods District Hospital (Other); Lakeridge Health Corporation (Other); North Bay General Hospital (Unknown); North York General Hospital (Other); Northumberland Hills Hospital (Unknown); Orillia Soldiers' Memorial Hospital (Unknown); Peterborough Regional Health Centre (Other); Sault Area Hospital (Other); Scarborough General Hospital (Other); Scarborough Grace Hospital (Unknown); Sudbury Regional Hospital (Unknown); Royal Victoria Hospital Of Barrie (Unknown); Michael Garron Hospital (Other); West Parry Sound Health Centre (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: OCCTKN
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2005-06

CONDITIONS: Ventilator Acquired Pneumonia; Catheter Related Blood Stream Infections; Pressure Ulcer Prophylaxis; DVT Prophylaxis; Restrictive Blood Transfusion Strategy; Daily Spontaeous Breathing Trials
Keywords: best practices, performance improvement, intensive care, measurement
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

INTERVENTIONS:
Behavioral: Focused knowledge translation strategies

SUMMARY:
The pragmatic issue at hand how to get physicians and nurses to use best practices… and how to measure consequences of their implementation. This is the science of "knowledge translation", which we are realizing is an "organic" entity. As part of our Critical Care Strategy our goal is to improve the quality and continuity of critical care within our health care system. Toward this goal we are implementing a program which links 16 Ontario hospitals through their critical care units in a Provincial Network.

ELIGIBILITY:
Inclusion Criteria:

* Cohort of hospitals with Intensive Care Units in Ontario

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-11; Study Completion 2007-09

PRIMARY OUTCOMES:
Relative risk of receiving best practices in the ICU.

SECONDARY OUTCOMES:
ICU length of stay
Barriers to best practice use in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: William J Sibbald, MD, MPH, Principal Investigator — Sunnybrook & Women's College Health Science Centre; Damon Scales, MD, MSc, Study Director — Sunnybrook & Women's College Health Sciences Centre
Locations (1):
- Sunnybrook & Women's College Health Science Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Scales DC, Dainty K, Hales B, Pinto R, Fowler RA, Adhikari NK, Zwarenstein M. A multifaceted intervention for quality improvement in a network of intensive care units: a cluster randomized trial. JAMA. 2011 Jan 26;305(4):363-72. doi: 10.1001/jama.2010.2000. Epub 2011 Jan 19. PMID 21248161